CLINICAL TRIAL: NCT02539576
Title: A Phase I, Open-label, Single-dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of Abacavir/Dolutegravir/Lamivudine Fixed-dose Combination Tablets in Healthy Japanese Subjects
Brief Title: Pharmacokinetics, Safety and Tolerability Study of Abacavir/ Dolutegravir/ Lamivudine Fixed-dose Combination Tablets in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 204662
Record Dates: First submitted 2015-08-20; First posted 2015-09-03 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: pharmacokinetics; Healthy subjects; Abacavir/dolutegravir/lamivudine; Japanese; Fixed-dose combination; safety
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABC/DTG/3TC FDC (Experimental): Each subject will receive treatment with a single oral dose of ABC 600 mg/DTG 50 mg/3TC 300 mg FDC tablet administered under the fasted state
  Interventions: Drug: ABC/DTG/3TC FDC tablet

INTERVENTIONS:
Drug: ABC/DTG/3TC FDC tablet — ABC/DTG/3TC FDC will be supplied as purple, biconvex, oval tablets debossed with "572 Trı" on one side and plain on the other side. A single dose, with a unit dose strength of 600 mg/50 mg/300 mg will be administered orally.

SUMMARY:
The abacavir (ABC)/dolutegravir (DTG)/lamivudine (3TC) 600 milligrams (mg)/50 mg/300 mg fixed-dose combination (FDC) tablet is currently approved in the United States (US) and Europe. Although the pharmacokinetics (PK), safety and tolerability of ABC/DTG/3TC FDC tablets have been extensively studied in subjects not of Japanese heritage, these parameters have not been exclusively assessed in Japanese subjects. To support the marketing application in Japan, this single-dose, open-label study will characterize the PK, safety and tolerability of ABC/DTG/3TC FDC tablet in adult Japanese healthy subjects. A maximum of 12 subjects will be enrolled such that approximately 10 evaluable subjects complete the study. The study will consist of a screening, treatment phase (single oral dose under the fasted state) and follow-up visit (within 7-14 days of the last PK sample collected). The total duration of the study for each subject will be approximately up to 48 days.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Japanese subjects who were born in Japan with 4 ethnic Japanese grand parents and must not have lived outside Japan for more than 10 years with being a Japanese passport holder (current or expired).
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, and laboratory tests.
* Subject values for haematology and chemistry within the normal range. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilograms (kg) (110 pounds [lbs]) for men and >=45 kg (99 lbs) for women and body mass index (BMI) within the range 18.5-31.0 kilogram per meter square (kg/m^2) (inclusive).
* Male or female

Females- A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine [according to the sites standard of practice] human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

1. Non-reproductive potential defined as: pre-menopausal females with one of the following: Documented tubal ligation Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion Hysterectomy Documented bilateral oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
2. Reproductive potential and agrees to follow one of the options listed below in the modified list of highly effective methods for avoiding pregnancy in females of reproductive potential (FRP) from 30 days prior to the first dose of study medication and until 2 weeks after dosing with study medication and completion of the follow-up visit.

The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Capable of giving signed informed consent as described in the protocol which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.
* Documentation that the subject is negative for the human leukocyte antigen (HLA) B*5701 allele.

Exclusion Criteria:

* Alanine aminotransferase (ALT) >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTcF >450 millisecond (msec)

NOTES:

The QT duration corrected for heart rate (QTc) is the QTcF machine-read or manually over-read.

The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial.

For purposes of data analysis, QT interval corrected for heart rate using Bazett's formula (QTcB), QTcF, another QT correction formula, or a composite of available values of QTc will be used as specified in the reporting and analysis plan (RAP).

* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and GlaxoSmithKline (GSK) medical monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One unit is equivalent to 12 gram (g) of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood product in excess of 500 mL within 56 days
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero (pre-dose) to time of last quantifiable concentration (AUC[0-t]) following a single oral dose administration of ABC/DTG/3TC 600 mg/ 50 mg/ 300 mg FDC tablet in healthy, adult Japanese subjects | Day 1: Pre-dose and at 30 minutes, 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h and 72 h post dose.
  Blood samples for PK analyses will be collected at pre-dose and 30 minutes, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post- dose.
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinity]) following a single oral dose administration of ABC/DTG/3TC 600 mg/ 50 mg/ 300 mg FDC tablet in healthy, adult Japanese subjects | Day 1: Pre-dose and at 30 minutes, 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h and 72 h post dose.
  Blood samples for PK analyses will be collected at pre-dose and 30 minutes, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post- dose.
Maximum observed plasma concentration (Cmax) following a single oral dose administration of ABC/DTG/3TC 600 mg/ 50 mg/ 300 mg FDC tablet in healthy, adult Japanese subjects | Day 1: Pre-dose and at 30 minutes, 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h and 72 h post dose.
  Blood samples for PK analyses will be collected at pre-dose and 30 minutes, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post- dose.
Time of occurrence of Cmax (tmax) following a single oral dose administration of ABC/DTG/3TC 600 mg/ 50 mg/ 300 mg FDC tablet in healthy, adult Japanese subjects | Day 1: Pre-dose and at 30 minutes, 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h and 72 h post dose.
  Blood samples for PK analyses will be collected at pre-dose and 30 minutes, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post- dose.
Concentration at 24 h after dose administration (C24) following a single oral dose administration of ABC/DTG/3TC 600 mg/ 50 mg/ 300 mg FDC tablet in healthy, adult Japanese subjects | Day 1: Pre-dose and at 30 minutes, 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h and 72 h post dose.
  Blood samples for PK analyses will be collected at pre-dose and 30 minutes, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post- dose.
Terminal phase half-time (t1/2) following a single oral dose administration of ABC/DTG/3TC 600 mg/ 50 mg/ 300 mg FDC tablet in healthy, adult Japanese subjects | Day 1: Pre-dose and at 30 minutes, 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h and 72 h post dose.
  Blood samples for PK analyses will be collected at pre-dose and 30 minutes, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post- dose.
Apparent clearance following oral dosing (CL/F) following a single oral dose administration of ABC/DTG/3TC 600 mg/ 50 mg/ 300 mg FDC tablet in healthy, adult Japanese subjects | Day 1: Pre-dose and at 30 minutes, 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h and 72 h post dose.
  Blood samples for PK analyses will be collected at pre-dose and 30 minutes, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post- dose.
Percentage of AUC(0-infinity) obtained by extrapolation (%AUCex) following a single oral dose administration of ABC/DTG/3TC 600 mg/ 50 mg/ 300 mg FDC tablet in healthy, adult Japanese subjects | Day 1: Pre-dose and at 30 minutes, 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h and 72 h post dose.
  Blood samples for PK analyses will be collected at pre-dose and 30 minutes, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post- dose.
Terminal phase rate constant (Lambda-z) following a single oral dose administration of ABC/DTG/3TC 600 mg/ 50 mg/ 300 mg FDC tablet in healthy, adult Japanese subjects | Day 1: Pre-dose and at 30 minutes, 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h and 72 h post dose.
  Blood samples for PK analyses will be collected at pre-dose and 30 minutes, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post- dose.

SECONDARY OUTCOMES:
Safety as assessed by the number of subjects with adverse events (AE) and serious adverse events (SAE) | From Day-1 up to follow-up (approx. Day 18)
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Absolute values for composite of clinical chemistry parameters as a safety measure | Day-1 and follow-up (approx. Day 18)
  Clinical chemistry parameters includes blood urea nitrogen, potassium, aspartate aminotransferase, total and direct bilirubin, creatinine, sodium, alanine aminotransferase, total protein, glucose, calcium, alkaline phosphatase and albumin
Change from baseline values for composite of clinical chemistry parameters as a safety measure | Day-1 and follow-up (approx. Day 18)
  Clinical chemistry parameters includes blood urea nitrogen, potassium, aspartate aminotransferase, total and direct bilirubin, creatinine, sodium, alanine aminotransferase, total protein, glucose, calcium, alkaline phosphatase and albumin
Urinalysis assessments | Day-1 and follow-up (approx. Day 18)
Safety as assessed by systolic and diastolic blood pressure measurements | Day-1, pre-dose and at 4 h, 24 h, 48 h post-dose, and follow-up (approx. Day 18)
Safety as assessed by pulse rate measurements | Day-1, pre-dose and at 4 h, 24 h, 48 h post-dose, and follow-up (approx. Day 18)
Safety as assessed by 12-lead electrocardiogram (ECG) | Day-1 and follow-up (approx. Day 18)
  Single 12-lead ECG will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT correction using Fridericia's Formula (QTcF) intervals.
Absolute values for composite of clinical haematology parameters as a safety measure | Day-1 and follow-up (approx. Day 18)
  Clinical haematology parameters includes platelet count, red blood cell count, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, neutrophils, lymphocytes, monocytes, eosinophils and basophils
Change from baseline values for composite of clinical haematology parameters as a safety measure | Day-1 and follow-up (approx. Day 18)
  Clinical haematology parameters includes platelet count, red blood cell count, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, neutrophils, lymphocytes, monocytes, eosinophils and basophils

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Glendale, California, United States